CLINICAL TRIAL: NCT01504373
Title: Regional Distribution Differences Between Neurally Adjusted Ventilatory Assist and Pressure Support Ventilation
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jordan Rettig, Associate, Critical Care Medicine, Boston Children's Hospital
Other Study IDs: 10070341
Record Dates: First submitted 2011-11-04; First posted 2012-01-05 (Estimated); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Respiratory Failure
Keywords: NAVA; neurally adjusted ventilatory support; lung injury; ventilation; lung volume distribution; oxygen cost of breathing
MeSH Terms: conditions — Respiratory Insufficiency; Lung Injury; Respiratory Aspiration | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NAVA-PSV: Subject will receive 4 hours of NAVA followed by 4 hours of PSV.
  Interventions: Device: Neurally Adjusted Ventilatory Assist (NAVA)
- PSV-NAVA: Subject will receive 4 hours of PSV followed by 4 hours of NAVA.
  Interventions: Device: Neurally Adjusted Ventilatory Assist (NAVA)

INTERVENTIONS:
Device: Neurally Adjusted Ventilatory Assist (NAVA) — Subjects will be placed in the NAVA mode of ventilation.

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) is an FDA approved mode of mechanical ventilation. This mode of ventilation is currently in routine use in adult, pediatric and neonatal intensive care units. The electrical activity of the diaphragm, the largest muscle used during inspiration, is measured. The ventilator triggers (synchronizes patient effort) and applies proportional assistance based on measured electrical activity of the diaphragm (Edi). This electrical activity is measured through a feeding tube that also has a multiple-array esophageal electrode in it. This mode of ventilation has been proven to be equivalent to pressure support ventilation (PSV). Theoretically, the breath-to-breath control offered by NAVA may not only trigger faster and synchronize better, but provide the support deemed appropriate by the central nervous center on demand. Traditionally in the intensive care unit (ICU), pressure support is applied to subject breathing spontaneously. Pressure is set to achieve a given tidal volume. The influence of changing lung compliance not only from the lung disease itself, but the interactions of the respiratory muscles can drastically change minute ventilation and contribute to hyper- or hypoventilation. These changes are typically found on assessment of end-tidal carbon dioxide (CO2), blood gas, or oxygen saturation (SpO2) monitoring; all of which are potentially preventable if we allowed the central nervous system to control the ventilator. NAVA may allow us to couple the central nervous system (neuro-coupling) with the ventilator to provide real-time proportional assistance, reduce work of breathing and apply physiologic breathing patterns.

ELIGIBILITY:
Inclusion Criteria:

* All intubated and mechanically ventilated patients in our intensive care units (ICUs) will be screened for the following inclusion criteria:

  1. Age: 1 month to 18 years.
  2. Mechanically ventilated for longer than 6 hours
  3. Either:

     1. Eligible for a spontaneous breathing mode of ventilation (not receiving chemical paralytics and has an appropriate spontaneous respiratory drive/rate given the size and condition of the patient) as determined by the team.

        or
     2. Currently in the pressure support ventilation (PSV) or neurally adjusted ventilatory assist (NAVA) mode of ventilation

Exclusion Criteria:

1. Patients in which a nasal gastric or oral gastric tube is contraindicated. Examples are but not limited to: s/p esophagus, tracheal surgery, bleeding disorders, facial trauma.
2. Uncuffed endotracheal tube (ETT)
3. Cervical-spine injury that prohibits rolling the patient for electrical impedance tomography (EIT) band placement.
4. Difficult airway
5. Congenital cyanotic heart defects
6. Positive end expiratory pressure (PEEP) > 15 cmH2O
7. Fractional inspired oxygen concentration (FIO2) > 0.8
8. Peak inspiratory pressure (PIP) > 30 cmH2O
9. Patients who are receiving chemical paralysis
10. History of prematurity (birth at post-conceptual age <37 weeks)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Regional distribution difference measured by electrical impedence tomography (EIT) | Change from baseline regional distribution of ventilation after the 4th hour and after 8th hour
  Regional distribution difference measured by EIT. Area and upper to lower lung volume ratios (as determined with EIT) will be the primary data analyzed. Global and regional filling of the lung will be compared during pressure support ventilation and neurally adjusted ventilatory assist.
Oxygen and metabolic cost of breathing | Change from baseline oxygen cost of breathing and carbon dioxide production after the 4th hour and after the 8th hour
  Oxygen consumption (VO2), carbon dioxide production (VCO2), respiratory quotient (RQ), and Work of breathing (VO2/time) will be measured and compared between baseline, pressure support ventilation (PSV), and neurally adjusted ventilatory assist (NAVA) within each patient. Percent change will be compared between control (PSV) and NAVA group.

SECONDARY OUTCOMES:
Oxygenation | Monitored/recorded continuously for duration of study (8 hours total)
  Oxygen saturation measured by pulse oxymetry (SpO2), SpO2/FiO2 ratio, non-invasive oxygen content (SpOC), and frequency of desaturations will be recorded continuously and compared between pressure support ventilation (PSV) and neurally adjusted ventilatory assist (NAVA). Although not a primary outcome measure of this study, oxygenation will allow us to further determine the safety of NAVA compared to PSV.
Lung mechanics | Monitored/recorded every 30 seconds for duration of study (8 hours total)
  Compliance, peak inspiratory pressures, positive end expiratory pressure, tidal volumes, inspired oxygen concentration, electrical activity of the diaphragm (Edi), specific Edi (ratio of tidal volume to Edi), will be measured in each patient during pressure support ventilation and neurally adjusted ventilatory assist.

CONTACTS AND LOCATIONS:
Overall Officials: John Arnold, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States